CLINICAL TRIAL: NCT02935088
Title: Practical Evaluation of Fractional Flow Reserve (FFR) and Its Associated Alternate Indices During Routine Clinical Procedures
Brief Title: PRESSUREwire Study
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: SJM-CIP-10136
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Results first posted 2020-02-07 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Coronary Artery Disease; Acute Coronary Syndrome
Keywords: FFR; Percutaneous coronary intervention
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fractional Flow Reserve — Measurement of physiologic parameters
  Other Names: PressureWire

SUMMARY:
The purpose of this study is to understand routine use of FFR (Fractional Flow Reserve) and alternate indices in clinical practice. This study will determine the use and clinical outcome of FFR-guided PCI in patients presenting with either stable coronary artery disease, or in patients presenting with Acute Coronary Syndrome (ACS) on culprit and non-culprit lesions as well as during index and secondary procedures.

DETAILED DESCRIPTION:
The purpose of this study is to understand routine use of FFR and alternate indices in clinical practice. This study will determine the use and clinical outcome of FFR-guided PCI in patients presenting with either stable coronary artery disease, or in patients presenting with Acute Coronary Syndrome (ACS) on culprit and non-culprit lesions as well as during index and secondary procedures.

The study will also collect data on the routine use of coronary physiologic measurements such as adenosine-induced hyperemia FFR, FFR by contrast-induced hyperemia,

ELIGIBILITY:
Inclusion Criteria:

* Patient is presenting with STEMI, NSTEMI, unstable angina, or stable coronary artery disease
* Patient is planned to have FFR performed or underwent a cardiac catheterization where FFR was performed for further PCI (Percutaneous Cardiac Intervention) consideration
* Patient signs and dates written informed consent
* Patient is eighteen years of age or older at the time of consent

Exclusion Criteria:

* Patient has extremely tortuous or calcified coronary arteries
* Patient with a patent coronary artery bypass graft to the target vessel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients where FFR has been performed or is planned to be performed for further evaluation of PCI procedures, as per physician clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 2217 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2019-03-22 (Actual); Study Completion 2019-03-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Berry, MD, Principal Investigator — University of Glasgow
Locations (71):
- United States (4):
  - Heart Center Research, LLC, Huntsville, Alabama
  - Orlando Health, Orlando, Florida
  - Atlanta VA Medical Center, Decatur, Georgia
  - Providence Everett Medical Center, Everett, Washington
- Austria (2):
  - Allgemeines Krankenhaus Linz, Linz
  - Krankenhaus Lainz, Vienna
- Canada (2):
  - London Health Sciences Centre, London
  - Hopital Sacre Coeur, Montreal
- Egypt (2):
  - Aswan Cardiac Center, Aswān
  - Al Dorrah Heart Care Hospital, Cairo
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Hospital, Tartu
- Germany (5):
  - Universitätsklinikum Aachen, Aachen
  - St.-Johannes-Hospital, Dortmund
  - Medizinische Einrichtungen der Universität Düsseldorf, Düsseldorf
  - Kliniken der Friedrich-Alexander-Universitat, Erlangen
  - Kliniken Villingen-Schwenningen, Villingen-Schwenningen
- Greece (2):
  - Alexandra General Hospital, Athens
  - University Hospital of Ioannina, Ioannina
- India (11):
  - Postgraduate Institute of Medical Education & Research, Chandigarh
  - Apollo Hospital, Chennai
  - The Madras Medical Mission, Chennai
  - Medanta - The Medicity Hospital, Gūrgaon
  - Fortis Escorts Hospital, Jaipur, Jaipur
  - Lisie Hospital, Kochi
  - Caritas Hospital, Kottayam
  - Sunshine Hospitals, Secunderabad
  - Ananthapuri Hospitals and Research Institute, Thiruvananthapuram
  - Sree Chitra Tirunal Institute for Medical Sciences and tech., Trivandrum
  - Christian Medical College & Hospital, Vellore
- Italy (6):
  - Ospedale Maggiore-Bellaria, Bologna
  - Centro Cardiologico Monzino, Milan
  - Policlinico di Modena, Modena
  - Azienda Ospedaliera Monaldi, Napoli
  - Policlinico Universitario A. Gemelli, Roma
  - Ospedale di Trento - P.O.Santa Chiara, Trento
- Japan (13):
  - Gifu Heart Center, Gifu
  - Tokyo Medical University Hachioji Medical Center, Hachiōji
  - Kansai Rosai Hospital, Hyōgo
  - Tenyoukai Central Hospital, Kagoshima
  - Yokosuka Kyosai Hospital, Kanagawa
  - Kanazawa Cardiovascular Hospital, Kanazawa
  - Gunma Prefectural Cardiovascular Center, Maebashi
  - Nishinomiya Watanabe Cardiovascular Center, Nishinomiya-shi
  - Sapporo Cardiovascular Clinic, Sapporo
  - Tohoku University Hospital, Sendai
  - Higashi Takarazuka Satoh Hospital, Takarazuka
  - Tsuchiura Kyodo General Hospital, Tsuchiura-shi
  - Yokohama City University Medical Center, Yokohama
- Netherlands (5):
  - VU Amsterdam, Amsterdam
  - Onze Lieve Vrouw Gasthuis, Amsterdam
  - Amphia Hospital, Breda
  - Catharina Ziekenhuis, Eindhoven
  - Haga Ziekenhuis Locatie Leyenburg, The Hague
- Portugal (4):
  - Hospital Garcia de Orta, EPE, Almada
  - Santa Maria Hospital, Lisbon
  - Hospital do Divino Espírito Santo, Ponta Delgada
  - Centro Hospitalar Vila Nova Gaia, Vila Nova de Gaia
- Saudi Arabia (2):
  - King Abdullah Medical City, Mecca
  - King Khalid University Hospital, Riyadh
- Spain (7):
  - Hospital de Basurto, Bilbao
  - Hospital Asistencial Universitario de Burgos, Burgos
  - Hospital Universitario Donostia, Donostia / San Sebastian
  - Complejo Hospitalario de Jaen, Jaén
  - Hospital Universitario Son Espases, Palma de Mallorca
  - Complejo Hospital Nuestra Señora de la Candelaria, Santa Cruz de Tenerife
  - Hospital Universitario Marqués de Valdecilla, Santander
- United Kingdom (4):
  - Golden Jubilee National Hospital, Clydebank
  - Kettering General Hospital, Kettering
  - Royal Free Hospital, London
  - St. Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schampaert E, Kumar G, Achenbach S, Galli S, Tanaka N, Teraphongphom T, Ginn G, Zhang Z, Somi S, Amoroso G, Brueren G, Krasnow J, Knaapen P, Berry C; PRESSUREwire Investigators. A global registry of fractional flow reserve (FFR)-guided management during routine care: Study design, baseline characteristics and outcomes of invasive management. Catheter Cardiovasc Interv. 2020 Oct 1;96(4):E423-E431. doi: 10.1002/ccd.28827. Epub 2020 Mar 14. PMID 32170905

RESULTS

PARTICIPANT FLOW:
Groups:
- FFR-guided PCI Patients: Patients presented with either stable coronary artery disease (CAD) or acute coronary syndrome (ACS) who is undergoing Fractional flow reserve (FFR)-guided percutaneous intervention (PCI) procedure
Period: Overall Study
Arm/Group | FFR-guided PCI Patients
Started (Subjects consented) | 2217
Completed | 2115
Not Completed | 102

BASELINE CHARACTERISTICS:
Groups:
- FFR-guided PCI Patients: Patients presented with either stable coronary artery disease (CAD) or acute coronary syndrome (ACS) who are undergoing fractional flow reserve (FFR)-guided Percutaneous intervention (PCI)
Arm/Group | FFR-guided PCI Patients
Number analyzed (Participants) | 2217
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 653
  Male | 1564
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 326
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 46
  White | 1681
  More than one race | 0
  Unknown or Not Reported | 162
Region of Enrollment [Number; unit: participants]
  United States | 250
  Japan | 165
  Egypt | 30
  United Kingdom | 176
  Portugal | 29
  Spain | 43
  India | 97
  Greece | 26
  Saudi Arabia | 56
  Canada | 57
  Austria | 39
  Netherlands | 785
  Italy | 138
  Germany | 295
  Estonia | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With 12 Month Clinical Outcomes (MACE) Major Adverse Cardiac Events by FFR Values and Resting Indices
Description: Major adverse cardiac events (MACE) is defined as a 12-month composite, including all cause death, documented non-fatal myocardial infarction, and unplanned hospitalization leading to urgent revascularization.
  Fisher Exact test will be performed to evaluate the association between 12-month MACE event and binary FFR variables respectively using the following FFR; Low FFR group (FFR ≤ 0.8) and high FFR group (FFR > 0.8).
Time Frame: 12 months
Population: The denominators used in the calculations of adverse event rates will be determined according to the analysis population excluding subjects who are lost to follow-up through given time point without events.
Measure: Count of Participants; unit: Participants
Groups:
- FFR <= 0.80: Patients who had an FFR <= 0.80
- FFR > 0.8: Patients who had an FFR > 0.80
Arm/Group | FFR <= 0.80 | FFR > 0.8
Number analyzed (Participants) | 794 | 1394
Participants
  MACE | 50 | 51
  Death | 19 | 30
  Myocardial infarction | 20 | 23
  Urgent revascularization | 23 | 17

2. Other Pre Specified Outcome: Correlation of Resting Indices With FFR Values
Description: Linear correlation will be used for continuous variables to examine agreement between FFR values and resting indices.
Time Frame: at time of procedure
Population: The number of participants and lesions analyzed were based on the number of participants underwent both FFR and Pd/Pa measurements for this Outcome Measure
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Lesion
Groups:
- FFR-guided PCI Patients (Lesion Level): Patients presented with either stable coronary artery disease (CAD) or acute coronary syndrome (ACS). The analysis is performed on lesion level
Arm/Group | FFR-guided PCI Patients (Lesion Level)
Number analyzed (Participants) | 1990
Number analyzed (Lesion) | 2644
correlation coefficient | 0.55

3. Other Pre Specified Outcome: Number of Subjects Who Had a Change in Treatment Plan When FFR is Used Compared to the Initial Decision Based on Angiography Alone
Description: Treatment decision was defined as "changed" if there is at least one decision change based on FFR for multiple lesions; if none of the decisions was changed for the multiple lesions, the treatment decision is defined as "unchanged".
Time Frame: at time of procedure
Measure: Count of Participants; unit: Participants
Groups:
- FFR-guided PCI Patients: Patients presented with either stable coronary artery disease (CAD) or acute coronary syndrome (ACS)
Arm/Group | FFR-guided PCI Patients
Number analyzed (Participants) | 2196
Participants | 763

4. Other Pre Specified Outcome: Number of Subjects With 12-Month Clinical Outcomes (MACE) Major Adverse Cardiac Events of Follow-up Subjects in Whom the Use of FFR Did Not Lead to a Change in Treatment Decision vs Subjects in Whom the Use of FFR Led to a Change in Treatment Decision
Description: Number of subjects with 12-Month Clinical Outcomes (MACE) Major Adverse Cardiac Events of Follow-up subjects in whom the use of FFR did not lead to a change in treatment decision vs subjects in whom the use of FFR led to a change in treatment decision.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Change in Treatment Plan Patients: The population who has a change in treatment plan post FFR
- No Change in Treatment Plan Patients: The population who has no change in treatment plan post FFR
Arm/Group | Change in Treatment Plan Patients | No Change in Treatment Plan Patients
Number analyzed (Participants) | 760 | 1428
Participants
  MACE | 33 | 68
  Death | 16 | 33
  Myocardial infarction | 10 | 22
  Urgent revascularization | 14 | 26

5. Other Pre Specified Outcome: Number of Subjects With 12-month Clinical Outcomes (MACE) by Other PressureWire-derived Indices (Contrast FFR)
Description: Number of subjects with 12-month clinical outcomes (MACE) by other PressureWire-derived indices (contrast FFR).
  Major adverse cardiac events (MACE) is defined as a 12-month composite, including all cause death, documented non-fatal myocardial infarction, and unplanned hospitalization leading to urgent revascularization.
Time Frame: 12 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Pd/Pa ≤ 0.92: Patients who had an Pd/Pa ≤ 0.92
- Pd/Pa > 0.92: Patients who had an Pd/Pa > 0.92
Arm/Group | Pd/Pa ≤ 0.92 | Pd/Pa > 0.92
Number analyzed (Participants) | 320 | 1684
Participants
  MACE | 28 | 67
  Death | 9 | 35
  Myocardial infarction | 13 | 20
  Urgent revascularization | 17 | 21

6. Other Pre Specified Outcome: Correlation of Other PressureWire-derived Index, Contrast FFR With FFR Values
Description: Linear correlation of FFR and contrast FFR (cFFR). Only subjects that had both FFR and cFFR were used in the analysis.
Time Frame: at time of procedure
Population: The number of participants and lesions analyzed were based on the number of participants underwent both FFR and cFFR measurements for this Outcome Measure
Measure: Number; unit: correlation coefficient
Units Other Than Participants: Lesion
Arm/Group | FFR-guided PCI Patients
Number analyzed (Participants) | 496
Number analyzed (Lesion) | 659
correlation coefficient | 0.77

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Event (AE): Any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device under study.
Arm/Group | FFR-guided PCI Patients
All-Cause Mortality (participants affected / at risk) | 50/2217
Serious Adverse Events (participants affected / at risk) | 107/2217
Other Adverse Events (participants affected / at risk) | 114/2217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFR-guided PCI Patients (N=2217)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorders (Cardiac disorders) | 71 (71) — MI, Chest Pain, Heart Failure
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (4)
General disorders (General disorders) | 10 (10)
Infections and infestations (Infections and infestations) | 4 (4)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) — Dissection
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Nervous system disorders (Nervous system disorders) | 3 (3)
Renal and urinary disorders (Renal and urinary disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Acute Aneurysm Abdominalis (Surgical and medical procedures) | 1 (1)
Vascular disorders (Vascular disorders) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FFR-guided PCI Patients (N=2217)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 (3)
Cardiac disorders (Cardiac disorders) | 77 (77) — MI, Chest Pain
Gastrointestinal disorders (Gastrointestinal disorders) | 4 (4)
General disorders (General disorders) | 10 (10)
Infections and infestations (Infections and infestations) | 4 (4)
Dissection (Injury, poisoning and procedural complications) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8)
Nervous system disorders (Nervous system disorders) | 3 (3)
Renal Failure (Renal and urinary disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Acute Aneurysm Abdominalis (Surgical and medical procedures) | 1 (1)
Vascular disorders (Vascular disorders) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT02935088/Prot_SAP_000.pdf